CLINICAL TRIAL: NCT03781960
Title: Phase II Trial of Abemaciclib and Nivolumab for Subjects With Hepatocellular Carcinoma
Brief Title: Abemaciclib and Nivolumab for Subjects With Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety letter from sponsor
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 35218
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — abemaciclib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abemaciclib & Nivolumab (Experimental): Subjects will receive abemaciclib monotherapy 150mg twice daily for seven days then will initiate nivolumab 480mg IV every 28 days while continuing twice daily abemaciclib.
  Interventions: Drug: Abemaciclib; Drug: Nivolumab

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib will be given at a dose of 150mg by mouth twice daily continuously for the duration of trial therapy.
  Other Names: Verzenio
Drug: Nivolumab — Nivolumab will be administered at a dose of 480mg IV every 28 days. Treatment with nivolumab will begin after an initial 7-day treatment period with abemaciclib monotherapy.
  Other Names: Opdivo

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of the combination of nivolumab and abemaciclib for the treatment of hepatocellular carcinoma. Other goals of this study are to learn about the side effects that this combination of drugs may cause and to learn more about how these drugs work by studying blood and tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have hepatocellular carcinoma (HCC) that is inoperable (where surgery is not indicated due to disease extent, co-morbidities, or other technical reasons)
2. Histologic confirmation of HCC is not required for screening but is required prior to initiation of study treatment. Subjects with hepatocholangiocarcinoma or cholangiocarcinoma are not eligible.
3. Tumor must be positive for retinoblastoma (RB) expression by immunohistochemistry
4. Age > 18 years and ability to understand and the willingness to sign a written informed consent document.
5. ECOG performance status of 0 or 1
6. Childs-Pugh score of <7
7. Life expectancy of at least 12 weeks
8. Must be able to swallow tablets
9. Must be willing to comply with protocol procedures (including completion of diaries and outcome measures)
10. Local or loco-regional therapy to the liver (i.e. surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed > 4 weeks prior to enrollment
11. Must be willing to undergo a pretreatment and on-treatment biopsy and have a tumor site that is accessible for core needle biopsy
12. Measurable or evaluable disease as defined by RECIST v. 1.1
13. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days of the first dose of abemaciclib (see Appendix A for definition of childbearing potential). Female subjects of childbearing potential must use an approved contraceptive method (detailed in Appendix A) for the duration of the study and an additional 3 weeks after the final dose of abemaciclib.
14. Subjects with hepatitis B must have an HBV viral load < 100 IU/mL by PCR during screening
15. Must have adequate organ and hematopoietic function as defined below:

Exclusion Criteria:

1. Any history of a serious medical or psychiatric condition that would prevent the subject from signing the informed consent form
2. Pregnant or breastfeeding
3. Use of any chemotherapy within 3 weeks prior to the first study treatment date
4. Use of any experimental therapy within 4 weeks or 5 half-lives, whichever is longer, prior to the first study treatment date
5. Use of radiation within 2 weeks prior to the first study treatment date (4 weeks if radiation to liver as per section 4.1)
6. Prior treatment with a CDK 4/6 inhibitor
7. Prior treatment with a PD-1 or PD-L1 inhibitor
8. Those who have not recovered from adverse events < Grade 1 from prior therapy, with the exceptions of alopecia of any grade or stable peripheral neuropathy < Grade 2
9. Subjects may not receive concomitant anticancer agents or radiation. Antiviral agents aimed at treating infectious hepatitis are permitted
10. History of or suspected hypersensitivity to nivolumab or abemaciclib
11. Uncontrolled ascites
12. Esophageal varices requiring treatment within the past 6 months (banding or medication)
13. Subjects with uncontrolled brain metastases. Subjects with brain metastases must have stable neurological status following local therapy (surgery or radiation) for at least 4 weeks prior to first study treatment and must be off of steroids related to the brain metastases.
14. Any concurrent condition requiring the continued or anticipated use of systemic steroids beyond physiologic replacement dosing (excluding non-systemic inhaled, topical skin, nasal, and/or ophthalmic corticosteroids). All other systemic corticosteroids above physiologic replacement dosing must be discontinued at least 4 weeks prior to first study treatment
15. Active drug or alcohol use or dependence as documented in the chart that, in the opinion of the investigator, would interfere with adherence to study requirements
16. Active bacterial or fungal infection requiring IV therapy at the start of protocol treatment
17. A second primary malignancy that, in the judgment of the investigator, may affect the interpretation of results
18. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint (e.g. interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea)
19. Personal history of ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest
20. Prior organ allograft or allogeneic bone marrow transplantation
21. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
22. Active autoimmune disease, except for vitiligo, type 1 diabetes mellitus, asthma, atopic dermatitis, or endocrinopathies manageable by hormone replacement; other autoimmune conditions may be allowable at the discretion of the Principal Investigator
23. Any other conditions judged by the investigator that would limit the evaluation of the subject
24. HIV positive by PCR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Karasic, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 met inclusion criteria and began treatment.
Period: Overall Study
Arm/Group | Abemaciclib & Nivolumab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abemaciclib & Nivolumab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate is determined by the percentage of participants on study attaining a partial or complete response as noted per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib & Nivolumab
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Progression-Free Survival
Description: Progression-Free survival is determined from the start of study treatment until the time of documented disease progression or death per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) and iRECIST criteria (guidelines for response criteria for use in trials testing immunotherapies)
Time Frame: From the start of study treatment until disease progression, death, whichever came first up to 2 years
Population: All subjects who received study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib & Nivolumab
Number analyzed (Participants) | 7
months | 2.1 [1.6 to 5.6]

3. Secondary Outcome: Duration of Response
Description: Time from the first recorded partial response or complete response (whichever comes first) defined Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; until disease progression or death
Time Frame: up to 2 years
Population: Subjects with objective response
Measure: Number; unit: months
Arm/Group | Abemaciclib & Nivolumab
Number analyzed (Participants) | 1
months | 10.2

4. Secondary Outcome: Overall Survival
Time Frame: From the start of treatment to death, due to any cause or last patient contact alive, assessed up to 2 years
Population: All subjects who received study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib & Nivolumab
Number analyzed (Participants) | 7
months | 7.9 [2.6 to 22.7]

ADVERSE EVENTS:
Time Frame: From the initiation of any study procedures until 30 days following the last administration of study treatment, up to 2 years.
Arm/Group | Abemaciclib & Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib & Nivolumab (N=7)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib & Nivolumab (N=7)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
bloating (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Edema Limbs (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nail Changes (Skin and subcutaneous tissue disorders) | 1 (1)
Palmer-plantar erthrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
AST Increased (Investigations) | 7 (7)
ALT Increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 7 (7)
Alkaline Phosphate Increased (Investigations) | 6 (6)
Platelet Count Decreased (Investigations) | 6 (6)
Creatinine increased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 7 (7)
Weight loss (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
WBC Decreased (Investigations) | 7 (7)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03781960/Prot_SAP_ICF_001.pdf